CLINICAL TRIAL: NCT02144701
Title: A Randomized Trial Testing a Probiotic Enteric Regimen for Easing Complications of Transplant (Randomized PERFECT Trial)
Brief Title: Lactobacillus Rhamnosus GG in Reducing Incidence of Graft-Versus-Host Disease in Patients Who Have Undergone Donor Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, RWJMS, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2012001625; NCI-2013-00094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2012001625 (Other: IRB number); P30CA072720 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus rhamnosus GG (Experimental): Patients receive Lactobacillus rhamnosus GG PO QD for 1 year.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG; Other: laboratory biomarker analysis was not performed because of no differences in the clinical outcomes
- No intervention (No Intervention): Patients receive no intervention.

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — Given PO
  Other Names: Culturelle; Gefilus; LGG
  Arms: Lactobacillus rhamnosus GG
Other: laboratory biomarker analysis was not performed because of no differences in the clinical outcomes — Correlative studies
  Arms: Lactobacillus rhamnosus GG

SUMMARY:
This randomized pilot clinical trial studies Lactobacillus rhamnosus GG in reducing incidence of graft-versus-host disease in patients who have undergone donor stem cell transplant. Lactobacillus rhamnosus GG may be effective at preventing for graft-versus-host disease caused by a donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if hematopoietic stem cell transplant (HSCT) patients treated with a probiotic (Lactobacillus GG [Lactobacillus rhamnosus GG])-containing diet compared to those not assigned to receive probiotic have a lower incidence of grade 1 upper gastrointestinal (GI) or grade 2-4 lower GI acute graft-versus-host disease (GVHD) (aGVHD) using Center for International Blood and Marrow Transplant Research (CIBMTR) scoring than those not prescribed a probiotic.

II. To determine if HSCT patients treated with a probiotic-containing diet compared to those not assigned to receive a probiotic have a: a) lower rate of organ-specific acute aGVHD (intestinal tract, skin, liver); b) lower rate of moderate or severe chronic GVHD (National Institutes of Health [NIH] consensus scoring) at 6 months and 1 year post transplant; c) shorter duration of immunosuppressive therapy (normalized for age and degree of human leukocyte antigen [HLA] match); d) lower rate of bacterial and/or opportunistic infection.

SECONDARY OBJECTIVES:

I. To determine if allogeneic hematopoietic stem cell patients treated with a probiotic compared to those not assigned to receive a probiotic have differences in: a) composition and proportion of the major gut bacterial phylotypes in stool (to be analyzed for changes pre- and post-initiation of probiotics and for association with development of aGVHD); b) measures of inflammation as assessed by cytokine or receptor production (interleukin [IL]-6, IL-8, tumor necrosis factor [TNF]-alpha, TNF-receptor 1, interferon-gamma, IL-2R, IL-10); c) qualitative measures of immune reconstitution as determined by sequential measurements of conventional T cells, regulatory T regulatory, B cells and natural killer (NK) cells; d) antibody class/subclass production; e) biomarkers associated with GVHD-elafin, regenerating islet-derived 3 alpha (Reg3a), suppressor of tumorigenicity-2 (ST2), hepatocyte growth factor (HGF); and/or urinary tryptophan metabolites; f) markers of gut barrier function including blood levels of endotoxin and microbial deoxyribonucleic acid (DNA).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive Lactobacillus rhamnosus GG orally (PO) once daily (QD) for 1 year.

ARM II: Patients receive no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign informed consent
* Undergoing allogeneic HSCT from a related or unrelated donor
* Hematopoietic engraftment as evidenced by recovery of the absolute neutrophil count to greater than 500/mm^3 for > 3 days without filgrastim (G-CSF) support and within 40 days of transplant (i.e. complete blood counts [CBCs] obtained 3 or more days apart while off of G-CSF must demonstrate an absolute neutrophil count > 500/mm^3); if absolute neutropenia is not achieved due to a non-myeloablative transplant, the patient can be enrolled on day +21 to +40
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Evidence of GVHD at the time of enrollment as assessed clinically
* Serum creatinine greater than 3.0
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3 times the upper limit of normal
* Total bilirubin greater than 2 times upper limit of normal
* Prior use of probiotics within 3 months prior to enrollment
* Inability to take medications by mouth
* Prior history of inflammatory bowel disease or other chronic diarrheal illness
* Prior history of hypersensitivity to milk proteins
* Active Clostridium difficile infection or on prophylactic or tapering antibiotics for Clostridium difficile infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 02/18/2013 and was closed to accrual on 04/22/2016.
Pre-assignment Details: We are reporting results on 33 eligible patients. 18 patients were deemed ineligible.
Groups:
- Lactobacillus Rhamnosus GG: Patients receive Lactobacillus rhamnosus GG PO QD for 1 year.
  Lactobacillus rhamnosus GG: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Lactobacillus Rhamnosus GG | no Intervention
Started | 22 | 11
Completed | 13 | 8
Not Completed | 9 | 3
Not completed — development of relapse, GVHD or death | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Lactobacillus Rhamnosus GG): Patients receive Lactobacillus rhamnosus GG PO QD for 1 year.
  Lactobacillus rhamnosus GG: Given PO
  laboratory biomarker analysis: Correlative studies
- Arm II (no Intervention): Patients receive no intervention.
- Total: Total of all reporting groups
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention) | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 7 | 26
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 18 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 16 | 8 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 21 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 20 | 11
Participants | 10 | 4

2. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 4
Participants | 10 | 4

3. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 4
Participants | 10 | 4

4. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 4
Participants | 10 | 4

5. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 4
Participants | 10 | 4

6. Primary Outcome: Rate of Grade 1 Upper GI and/or 2-4 Lower GI aGVHD Assessed Using CIBMTR Scoring
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 4
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of one year.
Arm/Group | Arm I (Lactobacillus Rhamnosus GG) | Arm II (no Intervention)
All-Cause Mortality (participants affected / at risk) | 4/21 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 0/21 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes